CLINICAL TRIAL: NCT00005315
Title: Psychosocial Factors and Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4078; 5P01HL047540 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2024-07-18 (Actual); Status verified 2008-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
Keywords: Ambulatory blood pressure monitoring; Masked hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Masked Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tru-SEQ mRNA sequencing has been performed for a subsample of the Masked Hypertension Study.
  Urine, serum, and plasma are in storage
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the role of psychosocial factors in the development of hypertension and cardiovascular disease.

To estimate the prevalence of masked hypertension and its potential role in the development of subclinical cardiovascular disease To compare the reliability of office blood pressure (BP), home BP and ambulatory BP, and their associations with subclinical cardiovascular disease

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

The studies had several interrelated themes. One was to explore the relationships between environmental stress and blood pressure over a range of time courses, with acute laboratory studies at one extreme, and long- term prospective studies at the other. The basic model of stress included three elements: the objective nature of the stressor, the individual's perception of it, and his or her physiological susceptibility. This model incorporated elements of the Karasek Job Strain model and the Frankenhaueser effort-distress model, with two components corresponding to demand and control. A third dimension was social support. These models were tested under both laboratory and field conditions. Blood pressure was the main dependent variable, together with structural changes in the heart and carotid arteries. Five projects were included. Project l evaluated the ability of ambulatory blood pressure, and blood pressure variability, to predict cardiovascular morbidity, and also included a cross-sectional study comparing the relationships between blood pressure and target organ damage in Black and white individuals. The hypothesis that white coat hypertension is a condition associated with lower risk than sustained hypertension was also tested. Project 2 (the Work Site Blood Pressure Study) prospectively evaluated the effects of job strain and social support on blood pressure and other outcome variables in a working population. Project 3 studied psychosocial and hormonal factors influencing diurnal variations of blood pressure in women, including the changes associated with menstruation and the menopause. Project 4 (the Masked Hypertension Study) assessed the prevalence of masked hypertension (normal BP in the clinic setting, but elevated BP in one's usual environment) and its association with subclinical cardiovascular disease (CVD); ~50% of the sample was re-evaluated an average of 6 years later. Project 5 (Improving the Detection of Hypertension) had repeat assessments of clinic BP, home BP and ambulatory BP in order to evaluate the test-retest reliability of each, and compare their associations with subclinical CVD.

The study was renewed in FY 1998, FY 2003 and in FY 2009 to continue follow-up and analysis.

ELIGIBILITY:
Employed screening blood pressure <=160/105 mmHg not taking antihypertensive medication no evidence of secondary hypertension no history of cardiovascular disease (myocardial infarction, stroke, heart failure, peripheral vascular disease).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants were recruited from 4 worksites and seen at one of two study sites.
Sampling Method: Non-Probability Sample
Enrollment: 893 (Actual)
Dates: Start 1993-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
24-hour ambulatory blood pressure | baseline and follow-up (50% of sample, an average of 6.5 years later)
left ventricular mass index | cross-sectional (baseline) and change (an average of 6.5 years later)
  by 2-D echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Schwartz, PhD, Principal Investigator — Columbia University

REFERENCES:
- [Background] Devereux RB, Pini R, Aurigemma GP, Roman MJ. Measurement of left ventricular mass: methodology and expertise. J Hypertens. 1997 Aug;15(8):801-9. doi: 10.1097/00004872-199715080-00002. PMID 9280201
- [Background] Devereux RB. Do antihypertensive drugs differ in their ability to regress left ventricular hypertrophy? Circulation. 1997 Apr 15;95(8):1983-5. doi: 10.1161/01.cir.95.8.1983. No abstract available. PMID 9133501
- [Background] Devereux RB, Agabiti-Rosei E, Dahlof B, Gosse P, Hahn RT, Okin PM, Roman MJ. Regression of left ventricular hypertrophy as a surrogate end-point for morbid events in hypertension treatment trials. J Hypertens Suppl. 1996 Sep;14(2):S95-101; discussion S101-2. doi: 10.1097/00004872-199609002-00018. PMID 8934385
- [Background] Roman MJ, Pickering TG, Schwartz JE, Pini R, Devereux RB. Relation of arterial structure and function to left ventricular geometric patterns in hypertensive adults. J Am Coll Cardiol. 1996 Sep;28(3):751-6. doi: 10.1016/0735-1097(96)00225-2. PMID 8772767
- [Background] Kim M, Roman MJ, Cavallini MC, Schwartz JE, Pickering TG, Devereux RB. Effect of hypertension on aortic root size and prevalence of aortic regurgitation. Hypertension. 1996 Jul;28(1):47-52. doi: 10.1161/01.hyp.28.1.47. PMID 8675263
- [Background] Cavallini MC, Roman MJ, Blank SG, Pini R, Pickering TG, Devereux RB. Association of the auscultatory gap with vascular disease in hypertensive patients. Ann Intern Med. 1996 May 15;124(10):877-83. doi: 10.7326/0003-4819-124-10-199605150-00003. PMID 8610916
- [Background] Saba PS, Roman MJ, Ganau A, Pini R, Jones EC, Pickering TG, Devereux RB. Relationship of effective arterial elastance to demographic and arterial characteristics in normotensive and hypertensive adults. J Hypertens. 1995 Sep;13(9):971-7. doi: 10.1097/00004872-199509000-00006. PMID 8586832
- [Background] James GD, Toledano T, Datz G, Pickering TG. Factors influencing the awake-sleep difference in ambulatory blood pressure: main effects and sex differences. J Hum Hypertens. 1995 Oct;9(10):821-6. PMID 8576898
- [Background] Gerin W, Pickering TG. Association between delayed recovery of blood pressure after acute mental stress and parental history of hypertension. J Hypertens. 1995 Jun;13(6):603-10. doi: 10.1097/00004872-199506000-00005. PMID 7594416
- [Background] Roman MJ, Pickering TG, Pini R, Schwartz JE, Devereux RB. Prevalence and determinants of cardiac and vascular hypertrophy in hypertension. Hypertension. 1995 Aug;26(2):369-73. doi: 10.1161/01.hyp.26.2.369. PMID 7635548
- [Background] Okin PM, Roman MJ, Devereux RB, Kligfield P. Electrocardiographic identification of increased left ventricular mass by simple voltage-duration products. J Am Coll Cardiol. 1995 Feb;25(2):417-23. doi: 10.1016/0735-1097(94)00371-v. PMID 7829796
- [Background] Palmieri V, de Simone G, Roman MJ, Schwartz JE, Pickering TG, Devereux RB. Ambulatory blood pressure and metabolic abnormalities in hypertensive subjects with inappropriately high left ventricular mass. Hypertension. 1999 Nov;34(5):1032-40. doi: 10.1161/01.hyp.34.5.1032. PMID 10567178
- [Background] Saba PS, Roman MJ, Longhini C, Scorzoni D, Pini R, Devereux RB, Ganau A. Carotid intimal-medial thickness and stiffness are not affected by hypercholesterolemia in uncomplicated essential hypertension. Arterioscler Thromb Vasc Biol. 1999 Nov;19(11):2788-94. doi: 10.1161/01.atv.19.11.2788. PMID 10559027
- [Background] Gerber LM, Schwartz JE, Schnall PL, Devereux RB, Warren K, Pickering TG. Effect of body weight changes on changes in ambulatory and standardized non-physician blood pressures over three years. Ann Epidemiol. 1999 Nov;9(8):489-97. doi: 10.1016/s1047-2797(99)00028-9. PMID 10549882
- [Background] Kario K, Schwartz JE, Pickering TG. Ambulatory physical activity as a determinant of diurnal blood pressure variation. Hypertension. 1999 Oct;34(4 Pt 1):685-91. doi: 10.1161/01.hyp.34.4.685. PMID 10523347
- [Background] Liu JE, Roman MJ, Pini R, Schwartz JE, Pickering TG, Devereux RB. Cardiac and arterial target organ damage in adults with elevated ambulatory and normal office blood pressure. Ann Intern Med. 1999 Oct 19;131(8):564-72. doi: 10.7326/0003-4819-131-8-199910190-00003. PMID 10523216
- [Background] Devereux RB, Okin PM, Roman MJ. Left ventricular hypertrophy as a surrogate end-point in hypertension. Clin Exp Hypertens. 1999 Jul-Aug;21(5-6):583-93. doi: 10.3109/10641969909060991. PMID 10423084
- [Background] Saba PS, Ganau A, Devereux RB, Pini R, Pickering TG, Roman MJ. Impact of arterial elastance as a measure of vascular load on left ventricular geometry in hypertension. J Hypertens. 1999 Jul;17(7):1007-15. doi: 10.1097/00004872-199917070-00018. PMID 10419075
- [Background] Bella JN, Roman MJ, Pini R, Schwartz JE, Pickering TG, Devereux RB. Assessment of arterial compliance by carotid midwall strain-stress relation in hypertension. Hypertension. 1999 Mar;33(3):793-9. doi: 10.1161/01.hyp.33.3.793. PMID 10082489
- [Background] Bella JN, Roman MJ, Pini R, Schwartz JE, Pickering TG, Devereux RB. Assessment of arterial compliance by carotid midwall strain-stress relation in normotensive adults. Hypertension. 1999 Mar;33(3):787-92. doi: 10.1161/01.hyp.33.3.787. PMID 10082488
- [Background] Schnall PL, Schwartz JE, Landsbergis PA, Warren K, Pickering TG. A longitudinal study of job strain and ambulatory blood pressure: results from a three-year follow-up. Psychosom Med. 1998 Nov-Dec;60(6):697-706. doi: 10.1097/00006842-199811000-00007. PMID 9847028
- [Background] Slotwiner DJ, Devereux RB, Schwartz JE, Pickering TG, de Simone G, Ganau A, Saba PS, Roman MJ. Relation of age to left ventricular function in clinically normal adults. Am J Cardiol. 1998 Sep 1;82(5):621-6. doi: 10.1016/s0002-9149(98)00390-7. PMID 9732891
- [Background] Devereux RB, Okin PM, Roman MJ. Pre-clinical cardiovascular disease and surrogate end-points in hypertension: does race influence target organ damage independent of blood pressure? Ethn Dis. 1998;8(2):138-48. PMID 9681280
- [Background] de Simone G, Devereux RB, Kimball TR, Mureddu GF, Roman MJ, Contaldo F, Daniels SR. Interaction between body size and cardiac workload: influence on left ventricular mass during body growth and adulthood. Hypertension. 1998 May;31(5):1077-82. doi: 10.1161/01.hyp.31.5.1077. PMID 9576117
- [Background] Devereux RB, de Simone G, Pickering TG, Schwartz JE, Roman MJ. Relation of left ventricular midwall function to cardiovascular risk factors and arterial structure and function. Hypertension. 1998 Apr;31(4):929-36. doi: 10.1161/01.hyp.31.4.929. PMID 9535417
- [Background] Schwartz JE, Stone AA. Strategies for analyzing ecological momentary assessment data. Health Psychol. 1998 Jan;17(1):6-16. doi: 10.1037//0278-6133.17.1.6. PMID 9459065
- [Background] Landsbergis PA, Schnall PL, Deitz DK, Warren K, Pickering TG, Schwartz JE. Job strain and health behaviors: results of a prospective study. Am J Health Promot. 1998 Mar-Apr;12(4):237-45. doi: 10.4278/0890-1171-12.4.237. PMID 10178616
- [Background] Devereux RB, de Simone G, Roman MJ. Relations of left ventricular geometry and function to prognosis in hypertension. Adv Exp Med Biol. 1997;432:1-12. doi: 10.1007/978-1-4615-5385-4_1. No abstract available. PMID 9433506
- [Background] Roman MJ, Pickering TG, Schwartz JE, Cavallini MC, Pini R, Devereux RB. Is the absence of a normal nocturnal fall in blood pressure (nondipping) associated with cardiovascular target organ damage? J Hypertens. 1997 Sep;15(9):969-78. doi: 10.1097/00004872-199715090-00007. PMID 9321744
- [Background] de Simone G, Devereux RB, Daniels SR, Mureddu G, Roman MJ, Kimball TR, Greco R, Witt S, Contaldo F. Stroke volume and cardiac output in normotensive children and adults. Assessment of relations with body size and impact of overweight. Circulation. 1997 Apr 1;95(7):1837-43. doi: 10.1161/01.cir.95.7.1837. PMID 9107171
- [Background] Belkic KL, Schnall PL, Landsbergis PA, Schwartz JE, Gerber LM, Baker D, Pickering TG. Hypertension at the workplace--an occult disease? The need for work site surveillance. Adv Psychosom Med. 2001;22:116-38. doi: 10.1159/000059280. No abstract available. PMID 11477935
- [Background] Devereux RB, Bella J, Boman K, Gerdts E, Nieminen MS, Rokkedal J, Papademetriou V, Wachtell K, Wright J, Paranicas M, Okin PM, Roman MJ, Smith G, Dahlof B. Echocardiographic left ventricular geometry in hypertensive patients with electrocardiographic left ventricular hypertrophy: The LIFE Study. Blood Press. 2001;10(2):74-82. doi: 10.1080/08037050152112050. PMID 11467763
- [Background] James GD, Bovbjerg DH. Age and perceived stress independently influence daily blood pressure levels and variation among women employed in wage jobs. Am J Hum Biol. 2001 Mar-Apr;13(2):268-74. doi: 10.1002/1520-6300(200102/03)13:23.0.CO;2-Z. PMID 11460873
- [Background] Devereux RB, Roman MJ, Palmieri V, Okin PM, Boman K, Gerdts E, Nieminen MS, Papademetriou V, Wachtell K, Dahlof B. Left ventricular wall stresses and wall stress-mass-heart rate products in hypertensive patients with electrocardiographic left ventricular hypertrophy: the LIFE study. Losartan Intervention For Endpoint reduction in hypertension. J Hypertens. 2000 Aug;18(8):1129-38. doi: 10.1097/00004872-200018080-00019. PMID 10954006
- [Background] Kario K, James GD, Marion R, Ahmed M, Pickering TG. The influence of work- and home-related stress on the levels and diurnal variation of ambulatory blood pressure and neurohumoral factors in employed women. Hypertens Res. 2002 Jul;25(4):499-506. doi: 10.1291/hypres.25.499. PMID 12358133
- [Background] Landsbergis PA, Schnall PL, Pickering TG, Schwartz JE. Validity and reliability of a work history questionnaire derived from the Job Content Questionnaire. J Occup Environ Med. 2002 Nov;44(11):1037-47. doi: 10.1097/00043764-200211000-00010. PMID 12448355
- [Background] Hoshide Y, Kario K, Schwartz JE, Hoshide S, Pickering TG, Shimada K. Incomplete benefit of antihypertensive therapy on stroke reduction in older hypertensives with abnormal nocturnal blood pressure dipping (extreme-dippers and reverse-dippers). Am J Hypertens. 2002 Oct;15(10 Pt 1):844-50. doi: 10.1016/s0895-7061(02)03020-0. PMID 12372670
- [Background] Kario K, Schwartz JE, Gerin W, Robayo N, Maceo E, Pickering TG. Psychological and physical stress-induced cardiovascular reactivity and diurnal blood pressure variation in women with different work shifts. Hypertens Res. 2002 Jul;25(4):543-51. doi: 10.1291/hypres.25.543. PMID 12358139
- [Background] Lipsky SI, Pickering TG, Gerin W. World Trade Center disaster effect on blood pressure. Blood Press Monit. 2002 Aug;7(4):249. doi: 10.1097/00126097-200208000-00008. No abstract available. PMID 12198342
- [Background] Gerber LM, Schwartz JE, Cedeno-Mero C, Warren K, Pickering TG. Association of urinary albumin concentration with casual and ambulatory blood pressure: a similar relationship in normotensive and hypertensive subjects. Blood Press Monit. 2001 Oct;6(5):245-51. doi: 10.1097/00126097-200110000-00004. PMID 12055419
- [Background] Kario K, Schwartz JE, Davidson KW, Pickering TG. Gender differences in associations of diurnal blood pressure variation, awake physical activity, and sleep quality with negative affect: the work site blood pressure study. Hypertension. 2001 Nov;38(5):997-1002. doi: 10.1161/hy1101.095009. PMID 11711488
- [Background] de Simone G, Devereux RB, Kimball TR, Roman MJ, Palmieri V, Celentano A, Daniels SR. Relation of heart rate to left ventricular dimensions in normotensive, normal-weight children, adolescents and adults. Ital Heart J. 2001 Aug;2(8):599-604. PMID 11577834
- [Background] Roman MJ, Pickering TG, Schwartz JE, Pini R, Devereux RB. Relation of blood pressure variability to carotid atherosclerosis and carotid artery and left ventricular hypertrophy. Arterioscler Thromb Vasc Biol. 2001 Sep;21(9):1507-11. doi: 10.1161/hq0901.095149. PMID 11557680
- [Background] Kario K, McEwen BS, Pickering TG. Disasters and the heart: a review of the effects of earthquake-induced stress on cardiovascular disease. Hypertens Res. 2003 May;26(5):355-67. doi: 10.1291/hypres.26.355. PMID 12887126
- [Background] Landsbergis PA, Schnall PL, Pickering TG, Warren K, Schwartz JE. Lower socioeconomic status among men in relation to the association between job strain and blood pressure. Scand J Work Environ Health. 2003 Jun;29(3):206-15. doi: 10.5271/sjweh.723. PMID 12828390
- [Background] Haas DC, Gerber LM, Shimbo D, Warren K, Pickering TG, Schwartz JE. A comparison of morning blood pressure surge in African Americans and whites. J Clin Hypertens (Greenwich). 2005 Apr;7(4):205-9; quiz 210-1. doi: 10.1111/j.1524-6175.2005.03503.x. PMID 15860959
- [Background] Haas DC, Davidson KW, Schwartz DJ, Rieckmann N, Roman MJ, Pickering TG, Gerin W, Schwartz JE. Depressive symptoms are independently predictive of carotid atherosclerosis. Am J Cardiol. 2005 Feb 15;95(4):547-50. doi: 10.1016/j.amjcard.2004.10.032. PMID 15695154
- [Background] Gerin W, Chaplin W, Schwartz JE, Holland J, Alter R, Wheeler R, Duong D, Pickering TG. Sustained blood pressure increase after an acute stressor: the effects of the 11 September 2001 attack on the New York City World Trade Center. J Hypertens. 2005 Feb;23(2):279-84. doi: 10.1097/00004872-200502000-00009. PMID 15662215
- [Background] de Simone G, Daniels SR, Kimball TR, Roman MJ, Romano C, Chinali M, Galderisi M, Devereux RB. Evaluation of concentric left ventricular geometry in humans: evidence for age-related systematic underestimation. Hypertension. 2005 Jan;45(1):64-8. doi: 10.1161/01.HYP.0000150108.37527.57. Epub 2004 Nov 22. PMID 15557389
- [Background] Devereux RB. Left ventricular mass and stroke. What is the connection? JAMA. 1994 Jul 6;272(1):71-2. No abstract available. PMID 8007085